CLINICAL TRIAL: NCT06743503
Title: An Exploratory, Open-label Study of UB-VV400 in Combination With Rapamycin in Relapsed or Refractory B-cell Malignancies
Brief Title: UB-VV400 in Combination With Rapamycin in Relapsed or Refractory B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UB-VV400CI001
Record Dates: First submitted 2024-12-10; First posted 2024-12-20 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Large B-cell Lymphoma
Keywords: UB-VV400; relapsed or refractory; Large B-cell Lymphoma
MeSH Terms: conditions — Recurrence | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Interventions: UB-VV400 with or without Rapamycin. Dosage and Administration:single dose of UB-VV400 intravenous injection at Day 1.
  For subjects receiving rapamycin, dosing should be planned to be initiated on Study Day 4 and continued for up to 60 days, as tolerated .
  Interventions: Genetic: UB-VV400; Drug: Rapamycin

INTERVENTIONS:
Genetic: UB-VV400 — UB-VV400 is a third-generation, self-inactivating (SIN), replication-incompetent, lentiviral vector (LVV) investigational drug product
Drug: Rapamycin — In DF Stage 2, Rapamycin will be given in combination with UB-VV400. For subjects receiving rapamycin, rapamycin dosing will be once daily with a planned start date of Day 4 (approximately 72 hours after the administration of UB-VV400) and continuing for up to 60 days, as tolerated.

SUMMARY:
This is an exploratory, open-label, investigator-initiated trial (IIT) of the safety, efficacy, and PK/Pd of UB-VV400 alone and in combination with rapamycin in adult subjects with R/R LBCL. LBCL will include subjects with aggressive lymphoma, defined as diffuse large B-cell lymphoma (DLBCL) not otherwise specified (NOS), including high-grade lymphoma (HGL) with double/triple hit DLBCL; transformed DLBCL (tDLBCL), including Richter's transformation; follicular lymphoma Grade 3B (FL3B); and primary mediastinal B-cell lymphoma (PMBCL). The study will include subjects who have had prior CD19-directed CAR T-cell exposure and subjects who are CAR T cell-naive. Clinical unmet need exists in both populations.

The objective of this study is to determine the MTD/MAD and following study of UB-VV400 administered alone and in combination with rapamycin. The dose-finding (DF) portion will evaluate the safety profile of UB-VV400 administered at various dose levels (DLs) alone (Stage 1) and in combination with rapamycin (Stage 2).

The dose-expansion (DE) portion will further optimize the dose and define the safety profile and preliminary efficacy of UB-VV400 alone and/or in combination with rapamycin. The study will use the Bayesian optimal interval (BOIN) design to allocate subjects to various DLs to minimize exposure to subtherapeutic DLs while maintaining appropriate safety parameters. DF will consist of 2 stages: Stage 1 DF aims to identify the MTD of UB-VV400 monotherapy, and Stage 2 DF aims to identify the MTD of UB-VV400 in combination with rapamycin. DF will be initiated in Stage 1 with UB-VV400 monotherapy, administered IV and starting at DL1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 at time of consent.
2. Provide voluntary written informed consent.
3. Relapsed/refractory disease for subjects that are either CAR T-naive or CAR T-exposed.
4. Measurable disease according to Lugano 2014 criteria.
5. No serious concomitant diseases or active/uncontrolled infections.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Cardiac function: left ventricular ejection fraction (LVEF) ≥ 40%.
8. Pulmonary function: pulse oximetry ≥ 90% on room air at rest.
9. Renal function: serum creatinine ≤ 1.5 × age-adjusted upper limit of normal (ULN) or creatinine clearance ≥ 45 mL/min.
10. Absolute lymphocyte count (ALC) ≥ 0.2×10^9/L.
11. Alanine aminotransferase (ALT) ≤ 2.5 × ULN, aspartate aminotransferase (AST) ≤ 2.5 × ULN, AND total bilirubin < 1.5 × ULN.
12. No ongoing coagulopathies requiring periodic replacement of clotting factors (eg, fresh frozen plasma, cryoprecipitate).
13. Women of childbearing potential must:

    1. Have 2 negative pregnancy tests verified (one negative serum beta human chorionic gonadotropin [β-hCG] at screening and another within 48 hours prior to treatment withUB-VV400).
    2. Commit to "true abstinence" from heterosexual intercourse or agree to use and complywith highly effective, uninterrupted contraception for 12 months after administration of UB-VV400 .
    3. Abstain from breastfeeding for 12 months following administration of UB-VV400.
14. Men with partners of childbearing potential must commit to "true abstinence" from heterosexual intercourse or agree to use a highly effective form of contraception duringheterosexual contact with a pregnant individual or any individual of childbearing potential for 12 months after administration of UB-VV400, regardless of past vasectomy.
15. Subjects must agree not to donate blood, organs, sperm/semen, and/or egg cells for use for at least 1 year following treatment with UB-VV400 alone or in combination with rapamycin. Insufficient data are available to define a duration of time sufficient to make a recommendation on when it is safe to donate any tissue; therefore, subjects should not donate any tissue after administration of UB-VV400.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Subjects with current isolated central nervous system (CNS) tumor involvement.
3. Subjects with a prior malignancy whose clinical course or management has the potential to interfere with the safety and/or efficacy evaluation of the clinical trial.
4. Prior treatment with any of the following: allogeneic bone marrow transplantation, gene therapy, or adoptive cell transfer of any kind except for CAR T-cell therapy.
5. Treatment with prior CD22-directed therapy except for UB-VV400.
6. History of or active human immunodeficiency virus (HIV).
7. Active hepatitis B (HepB) or hepatitis C (HepC).
8. For subjects receiving rapamycin: a. History of angioedema; b. Pneumonitis (Grade 3 or greater).
9. Ongoing Grade > 2 toxicities from the last line of anticancer therapy.
10. Use of the following:

    1. Therapeutic systemic doses of corticosteroids (defined as > 20 mg prednisone equivalent) within 72 hours before dosing with UB-VV400.
    2. Approved targeted therapies:

    i. Small molecules: within 3 half-lives before dosing with UB-VV400 (see package insert). ii. Antibodies: within 14 days before dosing with UB-VV400. iii. CAR T therapy: within 28 days before dosing with UB-VV400. c. Autologous stem cell transplant within 28 days before dosing with UB-VV400. d. Cytotoxic chemotherapy (eg, alkylators, anthracyclines) within 14 days before dosing with UB-VV400.

    e. Any experimental agent (ie, not approved for disease/indication or with accepted consensus guidelines recommendation) within 4 weeks before dosing with UB-VV400 unless progression has been documented and a minimum of 3 half-lives has elapsed.

    f. Any immune-suppressing agent within 28 days before dosing with UB-VV400 (eg, tacrolimus, mycophenolate mofetil, immunosuppressive antibodies such as anti-tumor necrosis factor [TNF]/IL-6).

    g. Radiation within 4 weeks before dosing with UB-VV400 (palliative radiation to a symptomatic lesion[s] is allowed if at least one additional, non-irradiated, measurable lesion remains present to assess response).

    h. Prophylactic treatment with short-acting oral antiretroviral medications within 7 days before UB-VV400 administration. Long-acting antiretroviral prophylaxis is not allowed within 2 years of UB-VV400 treatment.
11. Allergies to rapamycin or supportive medications required for CAR T-cell toxicity management (eg, tocilizumab).
12. Systemic autoimmune diseases or immunodeficiency diseases (except for well-controlled type I diabetes with hemoglobin A1C [HbA1c] less than 8% or well-controlled thyroid disease, as assessed by the treating physician).
13. Ongoing CNS diseases (eg, seizure disorder, tremor, history of cerebral vascular accident [CVA]/recurrent transient ischemic attack [TIA]) that would preclude evaluation of immune effector cell-associated neurotoxicity syndrome (ICANS).
14. Presence of uncontrolled angina or other acute uncontrolled heart disease. Myocardial infarction within the previous 6 months. New York Heart Association (NYHA) Class III or IV. History of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
15. Actively receiving treatment in other interventional clinical trials. Note: continued follow-up on previous trials is allowed for survivorship, but no further investigational agents or assessments will be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2028-05-21 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v5.0 | up to 24 months
  Type, frequency, and severity of adverse events (AEs) and laboratory abnormalities
Maximum tolerated dose (MTD) or maximum administered dose (MAD) of UB-VV400 alone and in combination with rapamycin. | up to 24 months

SECONDARY OUTCOMES:
Objective response rate (ORR) per the Investigator using the Lugano 2014 criteria. | up to 24 months

OTHER OUTCOMES:
Quantification of Immune cell subset frequencies (T/B/NK cells) | up to 24 months
Complete response (CR) rate, as determined by the Investigator using the Lugano 2014 criteria. | up to 24 months
Durability of response (DOR), the duration of response for subjects who acheived PR and CR as determined by the Investigator using the Lugano 2014 criteria. | up to 24 months
Progression-free survival (PFS) and Overall survival (OS). | up to 24 months
Quantification of plasma cytokines. | up to 24 months
Detection of integrated UB-VV400 transgene sequence and expression of CAR in peripheral blood. | up to 24 months
Maximum concentration (Cmax) of UB-VV400 particle and CAR-T cells. | up to 24 months
Time of maximum concentration (Tmax) of UB-VV400 particle and CAR-T cells. | up to 24 months
Area under the concentration versus time curve: UB-VV400 AUC0-7; CAR-T cell AUC0-28. | up to 24 months
Rate of incidence of anti-drug antibody, as determined by antibodies to UB-VV400 cocal glycoprotein (UB-VV400 pseudotyping) and anti-CD22 CAR (payload protein). | up to 24 months
Characterization of target antigen expression and biomarkers associated with immune cell infiltration and immunosuppression, as determined by CD22, CD4, CD8, FOXP3, CD56, CD3, CD20 expression. | up to 24 months
Analysis of correlation between CD22 expression frequency/levels and depth of response (PR or CR). | up to 24 months
Analysis of correlation between CD22 expression frequency/levels and the incidence rate and severity of AE. | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lei Fan, Principal Investigator — Department of Hematology, Jiangsu Province Hospital, the First Afﬁliated Hospital of Nanjing Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin

IPD SHARING:
Plan to Share IPD: No